CLINICAL TRIAL: NCT05656755
Title: The Effect of a Specific Training Based on Strengthening on Running Related-injuries in a Novice Runner Population: a Pilot Prospective Randomized Trial
Brief Title: Strengthening Running Program in Novice Runners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-502
Record Dates: First submitted 2022-11-17; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Runner's Knee
Keywords: Running; Running related injuries; strengthening program; prevention; performance
MeSH Terms: interventions — Resistance Training; Running

STUDY DESIGN:
Intervention Model Description: Randomised control trial (pilot study)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator were blinded for group distribution and randomisation. They also were the outcome assessor and were therefore kept blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strengthening running program (Experimental): The experimental group will undergo a specific running training based on leg strength training and interval running
  Interventions: Other: Strengthening; Other: Running
- Running program (Active Comparator): This running group will serve as control and will undergo a traditional running program composed of only running
  Interventions: Other: Running

INTERVENTIONS:
Other: Strengthening — The strengthening exercises were executed with the body weight without any additional weight and were composed of exercises like the squats, the lunges, the plank, and the mountain climbers
  Arms: strengthening running program
Other: Running — running for two supervised training sessions of one hour, and one free session of 30 minutes per week during 24 weeks

SUMMARY:
The objectives of the study are comparing the risk of injury and the running performance among novice runners with two different training programmes. The first programme has less running volume but more strengthening than the second one which is a normal running programme with no specific strengthening program.

This study will provide necessary information for a multicentric study to come. The information needed for this bigger study are the sample size, the attrition rate, the drop-out rate and the feasibility of the timeline.

DETAILED DESCRIPTION:
The objectives of the study are comparing the risk of injury and the running performance among novice runners with two different training programmes. The first programme has less running volume but more strengthening than the second one which is a normal running programme with no specific strengthening program.

Hypothesis: A training programme with less running but strengthening exercises based on interval technique and strength could have similar or better results regarding running related injuries and performance compared to a normal training programme.

The experimentation will take place in Louvain-la-Neuve in Belgium. Most of the common trainings will take place on the 400m outdoor track field of of the University. A sample of local university students will be drawned. The sex proportion of the participants should be representative of the population (non-runners population), thus 50/50. They will have to be non-runners in good and healthy condition. A non-runner is defined as someone who did not practice regular running at least twice a week for the last 6 months and could not perform a 10km at enrolment.

50 participants will take part in this experimentation. They will be randomized into 2 groups of 25. The investifator hypothesize that 40 participants will follow the study until the end.

ELIGIBILITY:
Inclusion Criteria:

1. they were between 18 and 30 years
2. matched our definition of novice runners
3. had not sustained a musculoskeletal injury in the past six months
4. agreed to subscribe to an online application and to report each running training on this platform.

A novice runner was defined as someone who has not been running more than once a week for more than six months. The participants were systematically excluded if they did not match the interval of age, were not considered as novice runners, i.e., ran twice or more times a week for more than six months

Exclusion Criteria:

* They were also excluded if they had sustained an injury in the last 6 months or suffered from any musculoskeletal or neurological disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic performance | at baseline
  aerobic performance testing using VAM-EVAL procedure
Aerobic performance | at 21 weeks of training
  aerobic performance testing using VAM-EVAL procedure

SECONDARY OUTCOMES:
Incidence of running related injuries | from baseline to 21weeks, up to 21 weeks total
  number of injuries due to running participation
drop-out | from baseline to 21weeks, up to 21 weeks total
  abandon from the running program for any reason except running related injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Irec/Nmsk, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No